CLINICAL TRIAL: NCT05899270
Title: Effect of 3D-printed Reconstruction Automated Matching System in Size Selection of Double-lumen Tube：a Prospective Double-blinded Randomised Controlled Trial
Brief Title: 3D-printed Reconstruction Automated Matching System Predicts Size of Double-lumen Tube: a Prospective Double-blinded Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Collaborators: Science and Technology Department of Sichuan Province (Other)
Responsible Party: Principal Investigator, Yihao Zhu, Clinical Professor, Sichuan Cancer Hospital and Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SCCHEC-02-2022-155
Record Dates: First submitted 2023-05-17; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Lung Cancer; Lung Diseases; Tracheal Intubation Morbidity; Throat Injury; Bronchus; Injury
MeSH Terms: conditions — Lung Neoplasms; Lung Diseases; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Participates recruited from Sichuan Cancer Hospital will randomized to 3D group and control group in 1:1 ratio via a random number list generated by a computer.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Two investigators performing intubation of DLT will be blinded to the intervention. All participates and researchers responsible for surgery, bronchoscopy assessment, follow-up, data management and analysis will also be blinded to the grouping.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D group (Experimental): In 3D group, the investigator will intubate using DLT chosen by an automatic comparison software for 3D reconstruction based on CT data (3DRACS).
  Interventions: Other: 3D reconstruction automatic matching system
- control group (Placebo Comparator): In control group, the size of DLT is based on patient's sex and weight and the height is used to guide the depth of DLT insertion.
  Interventions: Other: traditional method for selecting double lumen tube

INTERVENTIONS:
Other: 3D reconstruction automatic matching system — it is an automatic comparison software for 3D reconstruction based on CT data (3DRACS). It reconstructs the trachea and bronchus and compares them with the DLT, predicting the most suitable size and depth of the DLT for lung isolation.
  Arms: 3D group
Other: traditional method for selecting double lumen tube — In control group, the size of DLT is based on patient's sex and weight and the height is used to guide the depth of DLT insertion.
  Arms: control group

SUMMARY:
Lung isolation techniques are commonly used to facilitate surgical exposure and to provide single-lung ventilation for patients. We have developed an automatic comparison software for 3D reconstruction based on CT data (3DRACS). It reconstructs the trachea and bronchus and compares them with the DLT, predicting the most suitable size and depth of the DLT for lung isolation.The aim of this study was to compare whether the use of 3DRACS to select a DLT size compared to conventional empirical selection methods could improve incidence of DLT intubation success and reduce airway injury.

DETAILED DESCRIPTION:
Lung isolation techniques are commonly used to facilitate surgical exposure and to provide single-lung ventilation for patients undergoing various intra-thoracic procedures. Lung isolation is primarily accomplished with a double-lumen tube (DLT) or bronchial blocker. One published study showed that residents with limited experience had a 40% error rate in accurately placing a DLT. The accurate choice of the size of DLT is a prerequisite for good lung isolation.Currently, There is lack of proper objective criteria for selecting size of DLT. DLT size selection is estimated empirically using the patient's height and sex, and studies have shown that the size of DLT according CT images of the chest is more accurate than experience. we have developed an automatic comparison software for 3D reconstruction based on CT data (3DRACS). It reconstructs the trachea and bronchus and compares them with the DLT, predicting the most suitable size and depth of the DLT for lung isolation. The aim of this study was to compare whether the use of 3DRACS to select a DLT size compared to conventional empirical selection methods could improve incidence of DLT intubation success and reduce airway injury.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 75 years.
2. American Society of Anesthesiologists Physical Status (ASA-PS) I-III.
3. Planned to receive lung resection surgery during lung isolation techniques by using DLT.
4. Signed informed written consent.

Exclusion Criteria:

The participant experiences any of the following：

1. Spinal malformation,
2. Expected difficult airway
3. Tracheal stenosis
4. Tracheal tumor
5. Bronchial tumor
6. Distorted airway anatomy
7. Tumors of the mouth or neck

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of correct endobronchial intubation. | after intubation
  Conventional blindly endobronchial intubation is performed firstly and clinical verification was made by the same anesthesiologist, followed by the supervising anesthesiologist using a FOB to check DLT position and successful intubation was considered if the position was proper.

SECONDARY OUTCOMES:
Time to successful intubation | after intubation
  after completion of induction, the vocal cords are exposed using visual laryngoscopy and Cormack-Lehane grading is performed. The stopwatch is timed as soon as the cuff of DLT crosses the vocal cords and it stops when (1) intubating anesthesiologist consider the DLT is correctly positioned, (2) after a maximum of three attempts have been made, (3) the intubating anesthesiologist think DLT placed correctly is impossible. Each attempt is defined as returning the bronchial lumen of the DLT to the trachea and then attempting to reinsert it. If the DLT is unsuccessfully placed, the intubation will be performed under FOB guidance by the supervising anesthesiologist. This intubation time of supervising anesthesiologist is also counted as part of the successful intubation time.
Degree of pulmonary atrophy | after surgery begin
  it is a subjective score of 0-10 by the surgeon, ten mean very perfect, zero represent no pulmonary atrophy at all.
Grading of airway injury | When extubation
  an anesthesiologist over 10 years of FOB experience will assess tracheal and vocal cord related injuries from DLT intubation. Before DLT is prepared to extubation, FOB will be inserted into the bronchial lumen and the tracheal injury will be observed through the FOB along with DLT extubated. All images from the FOB assessment are saved as a video and it will be viewed are by another blinded endoscopist to assess the injury of vocal cords. The severity of tracheal injury was defined as follows: mild (redness, oedema, one to three speckled haemorrhagic lesions), moderate (over 3 mild lesions or one diffuse haemorrhagic lesion) and severe (more than 2 diffuse haemorrhagic lesions). With regard to the vocal cords, the types of lesions are classified as follows: (1) oedema, swelling of the mucosa; (2) petechiae, small red spots on the mucosa; (3) haematoma, bleeding into the mucosa.
Postoperative sore throat and hoarseness | At 1 hour and 24 hours after extubation
  sore throat is defined as persistent resting pain in the throat region, and throat pain scores were assessed by VAS score (0: no pain; 10: the most unbearable pain). Hoarseness is defined as a change in the quality of voice noted by the patient.
Oxygenation during one-lung ventilation | Intraoperative（from beginning of one lung ventilation to end），an average of 2 hours
  it is defined as the area under the curve of the SpO2/FiO2 ratio during OLV. The SpO2 and FiO2 values are automatically collected by the monitor at 30 second intervals and any abnormal data due to equipment or human error will be replaced with the previous correct data.
Account times of using FOB | During surgery (from induction to extubation), an average of 3 hour
  it was defined that FOB was inserted into the tracheal tube and then withdrawn from the tracheal tube from induction to extubation.

CONTACTS AND LOCATIONS:
Overall Officials: Yihao Zhu, master, Principal Investigator — department of anesthesiology, sichuan cancer hospital

IPD SHARING:
Plan to Share IPD: Yes
Data are available on reasonable request. The raw data are available from the corresponding author with applicable reason after publishing findings to a peer-reviewed journal.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The raw data are available from the corresponding author with applicable reason after publishing findings to a peer-reviewed journal.